CLINICAL TRIAL: NCT04737135
Title: Interstitial Myocardial Fibrosis in Repaired Tetralogy of Fallot: Assessment by Molecular and Imaging Biomarkers and Association With Adverse Events ( Myocardial FIbrosis in Repaired Tetralogy of FAllot- FIFA Study)
Brief Title: Myocardial FIbrosis in Repaired Tetralogy of FAllot- FIFA Study)
Acronym: FIFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PI 17/00149
Record Dates: First submitted 2021-01-20; First posted 2021-02-03 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect; Fallot Tetralogy
Keywords: Fallot Tetralogy; Myocardial fibrosis; T1-mapping; Collagen turnover biomarkers
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — serum, plasma and genomic DNA from blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with Tetralogy of Fallot
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Patients without intervention
  Other Names: Patients without intervention

SUMMARY:
This study aims to study the correlation between biomarkers of myocardial fibrosis (extracellular volume fraction calculated by cardiac magnetic resonance imaging (MRI) (T1-mapping) and levels of molecular biomarkers of fibrosis) and adverse events in a population of patients with repaired tetralogy of Fallot.

DETAILED DESCRIPTION:
The main causes of mortality in adults with repaired tetralogy of Fallot (TF) are sudden death and heart failure. Myocardial fibrosis has been linked to the appearance of arrhythmias and ventricular dysfunction in other patient populations, but this association is poorly studied in patients with TF, perhaps because research in congenital heart disease (CHD) requires multicenter studies, difficult to carry out. Interstitial myocardial fibrosis assessed by molecular and imaging biomarkers is associated with adverse events in patients with repaired Fallot tetralogy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with repaired tetralogy of Fallot or double outlet right ventricle Fallot type

Exclusion Criteria:

* Patients with pathologies that may interfere with the determination of the extracellular volume of myocardium (ischemic heart disease, storage diseases).
* Patients with pathologies that affect collagen metabolism (liver cirrhosis, stage ≥4 renal insufficiency, pulmonary fibrosis, metabolic bone disease, connective tissue diseases, active neoplasms, active treatment with corticosteroids and bone fractures or surgery in the previous 6 months).
* Pregnancy.
* Denial of informed consent.
* Patients with claustrophobia and pacemakers or defibrillators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with repaired tetralogy of Fallot or double outlet right ventricle Fallot type
Sampling Method: Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between myocardial fibrosis biomarkers and a composite of cardiac adverse events (cardiovascular death, sudden cardiac death, near-miss sudden death, supraventricular arrhythmias, ventricular arrhythmias, heart failure). | 4 years
  Myocardial fibrosis biomarkers: Cardiac Magnetic Resonance T1-mapping (extracellular volume fraction) and serum collagen turnover biomarkers (C-terminal propeptide of type I procollagen, C-terminal Telopeptide of type I Collagen, Matrix Metalloproteinase 1 and Tissue Inhibitor of Metalloproteinases-1)

SECONDARY OUTCOMES:
Correlation between myocardial fibrosis biomarkers and prior cardiac events (near-miss sudden death, supraventricular arrhythmias, ventricular arrhythmias and heart failure admissions). | up to time of reparative surgery
  Myocardial fibrosis biomarkers: Cardiac Magnetic Resonance T1-mapping (extracellular volume fraction) and serum collagen turnover biomarkers (C-terminal propeptide of type I procollagen, C-terminal Telopeptide of type I Collagen, Matrix Metalloproteinase 1 and Tissue Inhibitor of Metalloproteinases-1)
Correlation between myocardial fibrosis assessed by cardiac magnetic resonance (T1-mapping) and other cardiac magnetic resonance parameters (ventricular volumes, ejection fraction and strain). | Baseline
  Correlation of myocardial fibrosis assessed by cardiac magnetic resonance T1-mapping (extracellular volume fraction) and other cardiac magnetic resonance parameters (ventricular volumes, ejection fraction and strain).
Correlation between serum collagen turnover biomarkers and cardiac magnetic resonance parameters (ventricular volumes, ejection fraction and strain) | Baseline
  Correlation between serum collagen turnover biomarkers (C-terminal propeptide of type I procollagen, C-terminal Telopeptide of type I Collagen, Matrix Metalloproteinase 1 and Tissue Inhibitor of Metalloproteinases-1) and cardiac magnetic resonance parameters (ventricular volumes, ejection fraction and strain).
Correlation between myocardial fibrosis assessed by cardiac magnetic resonance (T1-mapping) and by serum collagen turnover biomarkers. | Baseline
  Correlation of myocardial fibrosis assessed by cardiac magnetic resonance T1-mapping (extracellular volume fraction) and by serum collagen turnover biomarkers (serum collagen turnover biomarkers (C-terminal propeptide of type I procollagen, C-terminal Telopeptide of type I Collagen, Matrix Metalloproteinase 1 and Tissue Inhibitor of Metalloproteinases-1).

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Universitari Valle de Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliver JM, Gallego P, Gonzalez AE, Garcia-Hamilton D, Avila P, Yotti R, Ferreira I, Fernandez-Aviles F. Risk factors for excess mortality in adults with congenital heart diseases. Eur Heart J. 2017 Apr 21;38(16):1233-1241. doi: 10.1093/eurheartj/ehw590. PMID 28077469
- [Background] Stefanescu Schmidt AC, DeFaria Yeh D, Tabtabai S, Kennedy KF, Yeh RW, Bhatt AB. National Trends in Hospitalizations of Adults With Tetralogy of Fallot. Am J Cardiol. 2016 Sep 15;118(6):906-911. doi: 10.1016/j.amjcard.2016.06.034. Epub 2016 Jun 27. PMID 27530825
- [Background] Puntmann VO, Peker E, Chandrashekhar Y, Nagel E. T1 Mapping in Characterizing Myocardial Disease: A Comprehensive Review. Circ Res. 2016 Jul 8;119(2):277-99. doi: 10.1161/CIRCRESAHA.116.307974. PMID 27390332
- [Background] Chen CA, Tseng WY, Wang JK, Chen SY, Ni YH, Huang KC, Ho YL, Chang CI, Chiu IS, Su MY, Yu HY, Lin MT, Lu CW, Wu MH. Circulating biomarkers of collagen type I metabolism mark the right ventricular fibrosis and adverse markers of clinical outcome in adults with repaired tetralogy of Fallot. Int J Cardiol. 2013 Sep 10;167(6):2963-8. doi: 10.1016/j.ijcard.2012.08.059. Epub 2012 Sep 19. PMID 22999338